CLINICAL TRIAL: NCT06090383
Title: Wearable and Deep Learning-Based Recognition of Real-World Movement Behavior of Adolescents With Cerebral Palsy: Feasibility and Discriminant Validity Study
Brief Title: Feasibility and Discriminant Validity of Monitoring Movement Behavior of Adolescents With Cerebral Palsy
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jan Christensen, Senior researcher, Rigshospitalet, Denmark
Other Study IDs: Sensor-H-22032100
Record Dates: First submitted 2023-10-09; First posted 2023-10-19 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Palsy (CP)
Keywords: Real-world; Movement Behavior; Adolescents; Cerebral Palsy; Wearables; Feasibility; Validity
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents with CP and typically developed adolescents.

SUMMARY:
A new artificial intelligence network has been developed to monitor real-world daytime and nighttime movement behavior of adolescents with cerebral palsy (CP). The network uses seven wearable sensors to recognize lying, sitting, and standing, as well as walking and movements of both arms and legs. This information can be useful for healthcare professionals to understand and influence change in movement behavior, leading to benefits for the health of adolescents with cerebral palsy. This study aims to examine the acceptability and technical dependability of monitoring the movement behavior of adolescents with cerebral palsy for 72 hours using wearable sensors. Additionally, the study aims to evaluate the network's ability to discriminate between control and individuals with CP, different subgroups of individuals with CP, as well as the incidence of sleep disturbance in the entire cohort.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a non-progressive disorder resulting from injuries or abnormalities in fetal or early infant brain development. According to registries from European countries, the condition affects 2-3 out of every 1000 live births. An individual with CP typically presents with motor development disorders that cause abnormal patterns of movement and posture due to impaired coordination of movements and muscle tone regulation. People with cerebral palsy can also have various other problems, including sensory and cognitive problems and sleep disturbances. These symptoms result in limitations in activity level and societal participation throughout the individual's life. Adolescents and even children as young as seven may experience a decline in motor ability, leading to changes in their movement behavior. Healthcare professionals rely on various observations and measurements performed in clinical and hospital settings to assess and treat individuals with CP. However, there is some uncertainty about whether these assessments truly reflect real-life movement behaviors, as using an impaired extremity in everyday life frequently deviates from its motor capacity. There is an absence of robust tools that capture daytime and nighttime movement behavior in real-world settings rather than in clinical or controlled environments. Hemiparesis is the most common marker of CP, making asymmetrical deficits a target for intensive interventions such as physical and occupational therapy. Yet, no clinical tools are available that document asymmetrical differences in the real world in children and adolescents with CP. An objective method to measure real-world movement patterns would allow therapists to identify individuals who need a more comprehensive evaluation and to target interventions and other management strategies more precisely. This would help children and adolescents with CP gain motor skills to maximize independence. Further, objectively observing individuals with CP in their daily lives is essential to gain insights into functional decline. It has been observed that children and adolescents with CP are more likely to experience sleep-related difficulties such as difficulty initiating sleep, frequent nocturnal awakenings, discomfort while in bed, and early morning awakenings. As sleep quality plays a vital role in health-related quality of life, it is crucial to have objective methods to evaluate and monitor potential sleep problems in a real-world context.

A deep-learning convolutional neural network has been modeled to recognize postures lying, sitting, and standing the activity of walking, and movements of the right and left extremities. The network uses accelerometer and gyroscope data from 7 wearable sensors. Testing of the network´s performance found that it surpasses human annotators in accurately classifying the movement behavior of healthy and typically developed adults. These findings are currently under review and have yet to be published. The present protocol details the methodology for assessing the feasibility of real-world movement behavior monitoring and the discriminant validity of the network in adolescents with CP and controls.

The feasibility evaluation examines the technology used, e.g., potential data loss and the credibility of data output, as well as user acceptance, e.g., sensor wear time and adverse events. The networks' discriminant ability will be assessed by the network's ability to differentiate between controls and CP severity, e.g., scores on the Gross Motor Functional Classification Scale - Expanded and revised (GMFCS-E&R), different types of CP, differently affected body parts of the participating adolescents with CP, as well as individuals who have and have not sleep problems in the entire cohort.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Cerebral Palsy at GMFCS-E&R levels I-V and typically developed without neurological impairment.
* Age range: 15-25 years
* Capable of providing informed consent or have a legal guardian who can provide consent on their behalf.

Exclusion Criteria:

* Adolescents without the capacity to provide informed consent when another young adult with the capacity can provide the same or similar data.
* Adolescents who have undergone musculoskeletal surgery or injury and have not resumed their normal movement behavior.
* Presence of skin wounds in areas where sensors are to be attached.

Ages: 15 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Primary care clinic and community sample
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Functional Classification Scale - Expanded and revised (GMFCS-E&R) | Day one
  The GMFCS-E&R is a classification system comprising five levels that aims to describe the gross motor function of children and adolescents with CP. This system considers five age bands; in this case, we use the 12-18-year-old age band. Individuals with CP are classified as level I when capable of walking without limitations, while those with non-ambulatory functions are classified as levels IV and V
Jenkins Sleep Evaluation Questionnaire (JSEQ) - Danish version | Day one
  The JSEQ evaluates the frequency and intensity of sleep difficulties in the past month. The questions pertain to difficulty falling asleep, frequent awakenings during the night, trouble remaining asleep, and subjective feelings of fatigue and sleepiness despite a typical night's rest. Respondents rate their experiences using a Likert-type scale, with the following response alternatives: not at all (1), 1 to 3 days (2), 4 to 7 days (3), 8 to 14 days (4), 15 to 21 days (5), and 22 to 28 days (6).

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Lorentzen, Prof., Principal Investigator — University of Copenhagen, Department of Neuroscience
Locations (1):
- University Hospital Copenhagen, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request

REFERENCES:
- [Background] Wimalasundera N, Stevenson VL. Cerebral palsy. Pract Neurol. 2016 Jun;16(3):184-94. doi: 10.1136/practneurol-2015-001184. Epub 2016 Feb 2. PMID 26837375
- [Background] Hanna SE, Rosenbaum PL, Bartlett DJ, Palisano RJ, Walter SD, Avery L, Russell DJ. Stability and decline in gross motor function among children and youth with cerebral palsy aged 2 to 21 years. Dev Med Child Neurol. 2009 Apr;51(4):295-302. doi: 10.1111/j.1469-8749.2008.03196.x. PMID 19391185
- [Background] Hulst RY, Gorter JW, Obeid J, Voorman JM, van Rijssen IM, Gerritsen A, Visser-Meily JMA, Pillen S, Verschuren O. Accelerometer-measured physical activity, sedentary behavior, and sleep in children with cerebral palsy and their adherence to the 24-hour activity guidelines. Dev Med Child Neurol. 2023 Mar;65(3):393-405. doi: 10.1111/dmcn.15338. Epub 2022 Jul 14. PMID 35833425
- [Background] Palisano RJ, Rosenbaum P, Bartlett D, Livingston MH. Content validity of the expanded and revised Gross Motor Function Classification System. Dev Med Child Neurol. 2008 Oct;50(10):744-50. doi: 10.1111/j.1469-8749.2008.03089.x. PMID 18834387

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/83/NCT06090383/SAP_000.pdf